CLINICAL TRIAL: NCT04421833
Title: Evaluation of the Effectiveness of the TOVERTAFEL System on Behavioral Disorders of People With Cognitive Disorders Hospitalized in Long-Term Care Units and in Reinforced Hosting Unit
Brief Title: Evaluation of the Effectiveness of the TOVERTAFEL System on Behavioral Disorders
Acronym: TOVERTAFEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL20_0145
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Behavioral Disorder
Keywords: dementia; non-drug intervention; apathy
MeSH Terms: conditions — Mental Disorders; Dementia; Lethargy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group starting with TOVERTAFEL activities (Active Comparator): Participants will benefit from TOVERTAFEL activities for 6 weeks then the usual animation techniques for 6 weeks with a week of wash-out between the two periods.
  Interventions: Behavioral: TOVERTAFEL; Behavioral: USUAL activities
- group ending with TOVERTAFEL activities (Sham Comparator): Participants will benefit from the usual animation techniques for 6 weeks then from TOVERTAFEL activities for 6 weeks with a week of wash-out between the two periods.
  Interventions: Behavioral: TOVERTAFEL; Behavioral: USUAL activities

INTERVENTIONS:
Behavioral: TOVERTAFEL — The TOVERTAFEL is a small box that can be attached to the ceiling. Inside the box is a high-quality projector, infrared sensors, a speaker, and a processor that work together to project games onto the table. Because the colored objects respond to the movements of the hands and arms, the residents can play with the light itself.
  The planned activities provide cognitive, social and physical stimulation through light projections and can all be used individually or in groups with the presence of a caregiver or facilitator. Sixteen play activities are offered.
Behavioral: USUAL activities — patients can participate in cooking workshops, cinema activities (screening of old films or documentaries on a large screen, in a "cozy" atmosphere), walks in the garden and the visit of a dog trained in assisted therapy by the animal.

SUMMARY:
The prevalence of behavioral disorders is high in patients living in an institutional environment or hospitalized in a long-term care unit. The consequences of these symptoms are not negligible with a faster cognitive decline and a significant impact on the life of the institution and of other patients when the disorders are pervasive and too difficult to manage for the healthcare teams.

Despite the daily attention paid to these disorders and their causes, especially the environmental ones, the teams are sometimes helpless, the teams are sometimes helpless today to fight against these symptoms, and their management thus constitutes a real challenge.

Non-drug interventions targeting this problem often require additional training, architectural installations (Snoezelen space) and / or are moderately effective. In order to offer a solution that can be used by everyone, that is transportable and based on new technologies, the TOVERTAFEL device was created.

These are interactive games projected onto a table using a ceiling projector. The light animations invite people to "play with the light" using arm or hand movements. These games stimulate residents' physical activity and encourage interactions between residents and with caregivers.

In this study, it is a question of evaluating the effectiveness of the TOVERTAFEL device on the frequent behavioral symptoms in dementia (agitation, ambulation, apathy, anxiety), the quality of life of the patients, as well as on psychotropic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 60 to 106.
* Patient living in one of the USLD or UHR participating in the project.
* Score greater than or equal to 9 for at least one of the following items in the NPI-ES: apathy, agitation, anxiety, depression, aberrant motor behavior.
* Presence of TNC according to the standardization and calibration of the MMSE.
* The patients recruited must have given themselves, or through a trusted person provided for in article L. 1111-6 of the Public Health Code, failing this, by the family, or, failing that, by a person having close and stable ties with the person concerned; for adults under guardianship: the guardian or legal representative, for adults under guardianship: the curator, their informed consent to this study which must be approved by the Personal Protection Committee (PPC) prior to its completion.

Exclusion Criteria:

* Unstable pathology whose nature can interfere with the evaluation variables
* Deafness or blindness which could compromise the patient's assessment or his participation in the animation sessions.

Ages: 60 Years to 106 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Behavioral and Psychological symptom dementia with Neuropsychiatric Inventory for Health Staff (NPI HS) after 6 weeks of intervention | 6 weeks
  The NPI-HS makes it possible to assess out of 12 each SPCD (delusions, hallucinations, agitation, depression, anxiety, elation, apathy, disinhibition, depression, aberrant motor behavior, sleep and appetite) according to its frequency (1: sometimes, 2: quite often, 3: frequently, 4; very frequently) and according to its severity (1: mild, 2: moderate, 3: significant). The score is calculated by multiplying the frequency and severity for each dimension and adding each of these sub-scores. The maximum score is 144. Responses to the NPI-ES are collected from the healthcare team by a psychologist before the start of the intervention, then at 6 weeks and 13 weeks of inclusion.

SECONDARY OUTCOMES:
Scores obtained before and after an intervention session on the Instantaneous Well-Being Assessment scale | before and after one intervention seance
  It is a visual analog scale allowing the patient to report on his state of well-being. In response to the question "How do you feel now / right now?" ", The patient will position their feeling of well-being by relying on pictograms representing simple facial expressions (joy, neutral and sadness) whose treatment is preserved late in the evolution of Alzheimer Disease. On the back, the positioning of the patient according to the pictograms is transcribed into a numerical value from 1 to 5. The answer "1" will correspond to the weakest feeling of well-being and the answer "5" to the feeling of the highest well-being.
Score obtained from the Caregiver Apathy Inventory after 6 weeks of intervention | 6 weeks
  The Caregiver Apathy Inventory collects information on the presence of apathy in patients with cerebral pathologies according to three dimensions: emotional dullness, loss of initiative, loss of interest. Each dimension is assessed by a caregiver according to its frequency (1: sometimes, 2: quite often, 3: frequently, 4; very frequently) and according to its severity (1: mild, 2: medium, 3: important). The score for each dimension is calculated by multiplying the frequency by the severity, obtaining a maximum score of 12. The total score of IA-S is obtained by adding the scores of the 3 dimensions obtaining a maximum score of 36.
Evolution of the consumption of psychotropic drugs before the start of the intervention | 6 weeks
  The evolution of the number of antidepressant, antipsychotic, anxiolytic and hypnotic drugs per patient will be compared according to the period (Tovertafel or usual animation techniques). For the patients concerned, the consumption of benzodiazepines translated into the administered dose equivalent to oxazepam will also be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital des Charpennes, Villeurbanne, France